CLINICAL TRIAL: NCT03879070
Title: Experimentation of an Ankle Mobilization Device for the Rehabilitation of Patients With Acquired Brain Injuries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: The National Research Council, Italy (Other Government); Regione Lombardia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIP599
Record Dates: First submitted 2019-03-13; First posted 2019-03-18 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: Ankle active and passive mobilization using an Ankle mobilization device
- Control group (No Intervention)

INTERVENTIONS:
Device: Ankle active and passive mobilization using an Ankle mobilization device — The treatment consists in 20 rehabilitation sessions, 5 times/week for 4 weeks. The device is capable of generating ankle dorsi/plantarflexion movements using two activation modes: passive and assistive. In the passive mode the device generates a movement pattern which the patient follows passively without exerting any force on the device. During the assistive mode, the device follows the active movement of the patient. During the intervention, these two modes will be alternated.
  Arms: Intervention group

SUMMARY:
The proposed clinical investigation plan is a randomized controlled pivotal study with 2 parallel groups, has a total duration of two years. For the study, 30 pediatric patients suffering from acquired brain injury will be recruited at the Scientific institute Eugenio Medea.

The primary aim of this study is to assess the clinical benefit of using an ankle mobilization device for the rehabilitation of pediatric patients with acquired brain injuries, on its clinical performance and its risks, and on its safety.

The efficacy of the treatment will be evaluated in terms of ankle range of motion (primary outcome). The effects of the treatment on musculoskeletal plasticity will be studied using an isokinetic machine and functional magnetic resonance imaging will provide information on variations of reactivity in the motor cortical network. Ease of use, safety and usability of the device will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Tetraplegic and hemiplegic acquired brain injury patients, within first month of injury.
* Spastic syndrome (ankle joint Modified Ashworth Scale > 1).

Exclusion Criteria:

* Pace maker or other contraindication to Magnetic Resonance Imaging scans.
* Other serious comorbidity.
* Behaviour and psychiatric disorders.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Passive range of motion of ankle dorsi-plantarflexion | Change from baseline after 4 weeks of treatment
  Measured with goniometer

SECONDARY OUTCOMES:
Ankle joint stiffness | Change from baseline after 4 weeks of treatment
  Device: isokinetic machine
Medical Research Council (MRC) Scale for Muscle Strength | Change from baseline after 4 weeks of treatment
  Scale for measuring Muscle Strength, range 0-5, higher is better.
Cerebral activation | Change from baseline after 4 weeks of treatment
  functional Magnetic Resonance blood oxygenation level dependent imaging
Time-Domain Near-Infrared Spectroscopy | Change from baseline after 4 weeks of treatment
  Blood oxygen saturation in muscles

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy